CLINICAL TRIAL: NCT06927609
Title: Effects of Kendall Exercises on Posture-Related Cervical Spondylosis
Brief Title: Kendall Exercises on Posture-Related Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/muhammad talha 02008
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cervical Spondylosis
Keywords: kendell exercise; Cervical spondylosis,; Postural abnormalities
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Kendall Exercises) (Experimental): Stretching of Cervical Extensors Strengthening Deep Cervical Flexors Strengthening Shoulder Retraction Stretching Pectoralis Muscle
  Interventions: Other: kendall exercises
- conventional therapy (Active Comparator): Cervical Traction Neck Isometric Exercises (Cervical flexors), Static Stretching (Cervical extensors) General Cervical Extension and Flexion Exercises Shoulder Shrugs
  Interventions: Other: Conventional therapy group

INTERVENTIONS:
Other: kendall exercises — Stretching of Cervical Extensors Strengthening Deep Cervical Flexors Strengthening Shoulder Retraction Stretching Pectoralis Muscle
  Arms: (Kendall Exercises)
Other: Conventional therapy group — Cervical Traction Neck Isometric Exercises (Cervical flexors), Static Stretching (Cervical extensors) General Cervical Extension and Flexion Exercises Shoulder Shrugs
  Arms: conventional therapy

SUMMARY:
This study evaluates the effectiveness of Kendall exercises in correcting postural deviations, such as forward head posture, associated with cervical spondylosis. By targeting muscle imbalances and improving alignment through stretching and strengthening protocols, the research aims to reduce symptoms, enhance cervical spine function, and promote postural health. Participants will undergo a four-week exercise intervention with pre- and post-assessments to determine the outcomes.

DETAILED DESCRIPTION:
This study investigates the impact of Kendall exercises on posture-related cervical spondylosis, a degenerative condition often linked to postural deviations like forward head posture (FHP). Prolonged poor posture, frequently exacerbated by activities such as excessive smartphone or computer use, leads to muscle imbalances, increased mechanical stress on the cervical spine, and degenerative changes in intervertebral discs and joints.

Kendall exercises are targeted therapeutic interventions designed to address muscle imbalances by strengthening weak muscles (e.g., deep cervical flexors) and stretching tight muscles (e.g., upper trapezius, pectoralis muscles). These exercises aim to restore proper alignment, reduce mechanical strain, and improve overall posture and cervical function.

Participants with posture-related cervical spondylosis will engage in a four-week exercise protocol involving specific Kendall exercises for cervical extensors, flexors, shoulder retraction, and chest muscles. Outcomes will be assessed using craniovertebral angle measurements, photographic analysis, and subjective pain/function scales. The study seeks to establish Kendall exercises as a non-invasive, effective intervention for managing cervical spondylosis by correcting postural deviations and mitigating associated symptoms

ELIGIBILITY:
Inclusion Criteria:

* • Already diagnosed patients of cervical radiculopathy confirmed by clinical examination and imaging

  * A patient with a Forward Head Posture (FHP) (CVA angle less the 48-50 degrees is defined as Forward head posture
  * Positive Spurling test
  * Numbness of the arm, fingers, or shoulder
  * Cervical Postural assessment showing asymmetry (radiographic Analysis, and Posture Observation)
  * Chronic symptoms ≥ 1 year
  * Pain and Stiffness which limited range of motion in the cervical spine (Flexion less than 60°) (Extension less than 73°) (Lateral Flexion less than 13°-23° Rotation less than 80°)
  * Pain: moderate to severe level (≥5 on NPRS)

Exclusion Criteria:

* • History of Recent trauma to the cervical spine

  * Any psychological condition
  * Any specific cause of cervical radiculopathy (e.g., metabolic diseases, rheumatoid arthritis, osteoporosis)
  * Central or peripheral neurological signs
  * History of spinal surgery.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4 weeks
  The Numeric Pain Rating Scale is an eleven-point pain impression scale: the patient rates pain from 0 (no aggravation) to 10 (most exceedingly terrible possible pain). Mild 1-3, Moderate 4-6, Severe 7-10. It has good test-retest reliability (r=.79-.96) in individuals with chronic pain and musculoskeletal pathology.
Range Of Motion: Goniometer | 4 weeks
  A goniometer is a tool used to measure joint angles and range of motion (ROM). The goniometer has high intra-rater and inter-rater reliability when used by trained professionals. Consistent measurement can be achieved with proper technique and positioning. It provides valid measurements of joint ROM when compared with other objective measures such as radiographic assessments.
craniovertebral angle (CVA) | 4 weeks
  The Craniovertebral Angle is one of the most reliable methods and common angles for evaluating the Forward head posture. It is the angle between a line drawn from the tragus of the ear to the C7 vertebra and a line drawn horizontally. A reduced CVA indicates a forward head posture.
Neck Disability Index (NDI) | 4 weeks
  The Neck Disability Index (NDI) is a widely used self-reported questionnaire that measures the patient's perceived disability due to neck pain. It consists of 10 items, each scoring from 0 to 5, covering various aspects such as pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Cronbach's alpha value for NDI was found to be .95 and this was statistically significant (p<.01).

CONTACTS AND LOCATIONS:
Overall Officials: Maria khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Batkhela, and Bahadur Khan, Rozi Khan Memorial Hospital, Malakand, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No